CLINICAL TRIAL: NCT03646214
Title: Oral Appliance Therapy for Improving Sleep Quality During Pregnancy: A Controlled Clinical Trial
Brief Title: Improving Sleep Quality During Pregnancy Using an Oral Appliance
Acronym: PREGNCCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Emet D. Schneiderman, PhD, Professor, Biomedical Sciences, Texas A&M University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2018-0048
Record Dates: First submitted 2018-06-27; First posted 2018-08-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Snoring; Sleep Fragmentation
MeSH Terms: conditions — Snoring; Sleep Deprivation | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor reading the sleep studies will have the treatment arm masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Midline traction oral appliance (Experimental): Subjects will wear the oral appliance nightly for 4 weeks. Must snore or have other evidence of sleep disordered breathing.
  Interventions: Device: Midline traction oral appliance
- Control (No Intervention): Subjects who do do not wish to wear the oral appliance will have their sleep monitored in parallel to the experimental subjects for 4 weeks.

INTERVENTIONS:
Device: Midline traction oral appliance — Device positions the mandible forward to open airway; device can be titrated to gradually advance the mandible.
  Other Names: MyTAP oral appliance; Mandibular advancement device
  Arms: Midline traction oral appliance

SUMMARY:
Many pregnant women suffer from poor sleep quality and snoring. Evidence shows an increasing association between (1) sleep disordered breathing and (2) maternal cardiovascular disease and in-hospital death. Snoring is a variant of obstructive sleep apnea (OSA) and OSA during pregnancy is associated with higher risks for cesarean delivery, gestational hypertension, preeclampsia and preterm delivery. It may also impact fetal outcomes negatively. The purpose of this study is to determine whether sleep quality can be improved in pregnant women who snore by means of an oral appliance that opens the airway. Sleep quality is evaluated objectively using an un-intrusive home sleep test system.

DETAILED DESCRIPTION:
As many as 20 percent of women suffer from snoring and poor sleep quality while pregnant. The purpose of this study is to determine whether sleep can be improved in pregnant women who snore by means of a midline traction oral appliance (OA) that opens the airway. This is an interventional study to objectively evaluate OA therapy on breathing during sleep as well as its effect on sleep quality. Pregnant women from all trimesters will be recruited. Each subject is expected to participate in the study for at least five (5) consecutive weeks. Home sleep recordings will be collected at three time points: T0 - Baseline prior to OA use for two consecutive nights; T1- first two consecutive nights wearing the OA; T2 - for two consecutive nights after 4 weeks of appliance use. In addition to the sleep studies performed at each of these time points, subjects will also complete several brief surveys. All participants will be given the opportunity to use their OAs after the 4 week period, and have their sleep recorded at 8 week intervals through the remainder of their pregnancies. Participants will get to keep and use their OAs after the study.

Pregnant women who snore (or otherwise have poor sleep), may qualify to participate in this study. Those who do not want to wear an oral appliance, but are interested in learning about sleep quality while pregnant, may also qualify to participate as a control subject.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant adults who snore
* At least 8 teeth per arch
* Mallampati score from I to II
* Palatine tonsils grade 0,1 or 2
* Capable of giving verbal and written informed consent
* Able to apply the sleep recorder and the oral appliance.

Exclusion Criteria:

* Pregnant > 32 weeks
* Uncontrolled serious health issues
* Cardiovascular or cardiac rhythm disorders
* Pharmacological dependency
* Concomitant use of hypnotic agents or other sleep aids, nicotine or alcohol
* Ongoing temporomandibular joint disorders
* Loose teeth or periodontal disease
* History of uvulopalatopharyngoplasty (UPPP)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of stable to unstable sleep from CPC | Two nights of sleep recordings at each of 3 time point over 5 weeks.
  Ratio of stable to unstable sleep based on cardiopulmonary coupling analysis.

SECONDARY OUTCOMES:
Number of snores per hour of sleep | At each of 3 time points over 5 weeks
  Number of snores and snore index (#snores/hour of sleep)
Pittsburgh Sleep Quality Index (PSQI) | At baseline and after 5 weeks
  Self reported measures concerning sleep over a 1-month period; overall score ranging from 0 to 21; Scores >7 suggests poor sleep quality.
Insomnia Sleep Questionnaire (ISQ) | At baseline and after 5 weeks
  A screening tool used to guide in the clinical evaluation of insomnia; Scores 3, 4 or 5 to two or more items suggests significant daytime impairment and further evaluation of insomnia.
Hamilton Depression Rating Scale (HDRS) | At baseline and after 5 weeks
  Used to provide an indication of depression, and as a guide to evaluate recovery; Higher scores = depression severity. Score >20 suggests depression severity.
Fatigue Severity Scale (FSS) | At baseline and after 5 weeks
  9-item scale which measures the severity of fatigue and its effect on a person's activities; and lifestyle. Higher scores = greater fatigue severity. Minimum score = 9; Maximum score = 63.

CONTACTS AND LOCATIONS:
Overall Officials: Emet D Schneiderman, PhD, Principal Investigator — Texas A&M University College of Dentistry; Preetam J Schramm, PhD, Principal Investigator — Texas A&M University College of Dentistry
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No